CLINICAL TRIAL: NCT04479839
Title: Senior Atending Anesthesiologist
Brief Title: Point of Care Ultrasound to Confirm Endotracheal Tube Cuff Position in Relationship to the Cricoid in Pediatric Population.
Status: Completed | Type: Observational
Sponsor: Sidra Medicine (Other)
Responsible Party: Principal Investigator, Tariq Wani, Senior attending, Sidra Medicine
Other Study IDs: 1570971
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Endotracheal Tube; Cricoid Cartilage; Ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Microcuff ETT: Patients intubated with microcuff ETT
  Interventions: Diagnostic Test: Ultrasound of the airway
- Non-microcuff ett: Patients intubated with regular ETT
  Interventions: Diagnostic Test: Ultrasound of the airway

INTERVENTIONS:
Diagnostic Test: Ultrasound of the airway — Placing ultrasound on the neck after intubation

SUMMARY:
Anatomically, the infra-glottic area (subglottis) and the cricoid ring are the narrowest part of the larynx. In order to limit the incidence of damage related to mucosal pressure injuries from the presence of an endotracheal tube (ETT), the cuff of the ETT should lie below the cricoid in children. Previously, no clinical or imaging method has been used in real time at the bedside to determine the exact location of the ETT cuff after endotracheal intubation. Point-of-care ultrasound (POCUS) may provide an option for a safe and rapid means of visualizing the cuff of the ETT and its relationship to the cricoid ring in real-time thereby allowing ideal ETT positioning.

DETAILED DESCRIPTION:
Airway below vocal cords until the distal end of the cricoid referred to as subglottis or infraglottis is considered to be the narrowest part of the airway. An optimal endotracheal tube (ETT) placement with cuffed ETT is to ensure the cuff position below the cricoid ring (cuff free glottis): as well have sufficient distance between ETT tip and carina. Various modalities including clinical examination, ETCO2, imaging (X-ray and ultrasound) are routinely used to verify the position and the tip of the ETT in the airway, however verification of the cuff position remains obscure.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing general anesthesia requiring endotracheal intubation

Exclusion Criteria:

* Patients with any anatomical airway deformity or mass

Ages: 1 Day to 71 Months | Sex: All
Age Groups: Child
Study Population: 80 children from birth to 7 years, scheduled for the surgery requiring endotracheal intubation
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Visualize the saline-filled cuff of the endotracheal tube | 3 months
  The primary objective was to visualize the saline-filled cuff of the endotracheal tube in relation to the cricoid and tracheal rings

CONTACTS AND LOCATIONS:
Overall Officials: Tariq Wani, Principal Investigator — Attending physician
Locations (1):
- Sidra Medicine, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No